CLINICAL TRIAL: NCT00765089
Title: Bipolar Radiofrequency Ablation -Role in Prevention of Postoperative Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Lawrence Wei, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0508144
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Postoperative Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulmonary Vein isolation (Experimental): Patients in this arm will receive pulmonary vein isolation during surgery
  Interventions: Procedure: Isolation of pulmonary veins with Bipolar radiofrequency ablation
- Standard of care (No Intervention): Subjects in this arm will receive standard of care and no pulmonary vein isolation

INTERVENTIONS:
Procedure: Isolation of pulmonary veins with Bipolar radiofrequency ablation
  Arms: Pulmonary Vein isolation

SUMMARY:
Atrial Fibrillation (AF) is one of the most common postoperative complications after coronary artery bypass grafting (CABG). Postoperative AF produces a substantial impact on hospital resources with an estimated annual expenditure of over $1 billion. This includes the cost of pharmacological treatment and the cost of the increased length of stay. The incidence of AF is about 30-40% in CABG patients and increases with age of the patient. As the average age of the patient that undergoes CABG surgery is increasing, it is critical to find a way to prevent or reduce the incidence of this complication.

We propose a prospective, randomized, controlled study to determine the role of pulmonary vein isolation by bipolar ablation in the prevention or reduction of postoperative AF. The block- randomization plan will be used to maintain balance of the study and control arms throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who require an isolated elective CABG surgery on CPB.
2. Both male and female patients of age 18 years to 90 years.

Exclusion Criteria:

1. Pre existing atrial fibrillation or history of previous atrial fibrillation.
2. Inability to provide informed consent.
3. Pregnant or nursing patients.
4. Reoperative sternotomy
5. Emergency CABG surgery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Reduced incidence of Postoperative Atrial fibrillation | 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States